CLINICAL TRIAL: NCT04553484
Title: Measuring Cardiovascular Performance and Blood Flow Using Common But Never Compared Methods.
Status: Completed | Type: Observational
Sponsor: Semler Scientific (Industry)
Responsible Party: Sponsor
Other Study IDs: 35-0102
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: D012039; D001775

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All subjects enrolled: The feasibility of conducting all three tests, echocardiography (Echo), Brain Natriuretic Peptide (BNP) and volume plethysmography (VP), on all subjects met the enrollment criteria.
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Measuring Cardiovascular Performance Using Common Methods in subjects.

DETAILED DESCRIPTION:
This study will conduct measurements of cardiovascular performance by echocardiography (Echo), Brain Natriuretic Peptide (BNP) blood serum levels and blood flow by volume plethysmography (VP) in subjects who meet the AHA/ACC criteria for screening for peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* At least 50 Patients from New York Heart Association (NYHA) Class 1 (One or more AHA Risk Factors, asymptomatic), ≤75% (36) Male, ≥25% (12) Female
* At least 50 Patients from NYHA Class 2 (symptomatic), ≤75% (36) Male, ≥25% (12) Female

Exclusion Criteria:

* Subjects on mechanical ventilation.
* Subjects who require decisions by a medical power of attorney.
* Subjects unable to safely perform forced expiration.
* Subjects with known technically difficult (TDS) trans-thoracic echocardiographic windows.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 Years and older Female and Male
Sampling Method: Non-Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Kermode, Study Director — Semler Scientific
Locations (4):
- United States (4):
  - Middle Georgia Heart and Vascular Center, Macon, Georgia
  - Integrated Cardiology Group, LLC, d/b/a Bryan Heart, Lincoln, Nebraska
  - JF Southwest Heart Clinic, P.A., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Protocol was amended to include measurement of Brain Natriuretic Peptide (BNP) later in the study.
Groups:
- All Subjects Enrolled.: 1 day for the collection of the test results of the 657 participants was performed for Echocardiography and Volume plethysmography tests. And 1 day for the collection of Brain Natriuretic peptide (BNP) tests results of 236 participants was conducted.
Period: Overall Study
Arm/Group | All Subjects Enrolled.
Started | 657
Completed | 657 (The Protocol was amended to include measurement of Brain Natriuretic Peptide (BNP). Of the 657 participants, 236 had BNP measured.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Protocol was amended to include measurement BNP participants. 657 participants had Echo and VP, while 236 of the same 657 group of participants also had BNP measurement.
Groups:
- Measuring Cardiovascular Performance and Blood Flow.: Echocardiography (Echo), Brain Natriuretic Peptide (BNP), and volume plethysmography (VP) were performed in human subjects.
Arm/Group | Measuring Cardiovascular Performance and Blood Flow.
Number analyzed (Participants) | 657
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Protocol was amended to include 236 participants for the measurement of Brain Natriuretic Peptide (BNP).
  years | 61.5 (11.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 379
  Female | 276
  Not Recorded | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 657

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Performing Echo, BNP, and VP on Human Subjects.
Description: The feasibility of performing three common tests, Echocardiography (Echo), Brain Natriuretic Peptide (BNP) and volume plethysmography (VP), in the same subject was assessed. Each of the 657 participants were submitted to a brief non-invasive blood flow and cardiac performance test (plethysmography (VP) and Echocardiography (Echo)). Each of the 236 participants were subject to blood drawn test, Brain Natriuretic Peptide (BNP).
Time Frame: Baseline
Population: All subjects could safely do the Echo and VP tests, and after the protocol was amended, 100% of subjects could safely do the BNP as well. The quality of the test results was not assessed in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Echo, Volume Plethysmography: All subjects could safely do the Echocardiography (Echo) and volume plethysmography (VP) tests, and after the protocol was amended, 100% of subjects could safely do the Brain Natriuretic Peptide (BNP) as well. The quality of the test results was not assessed in this study.
- Brain Natriuretic Peptide (BNP): 236 subjects of the 657 subjects could safely do the Brain Natriuretic Peptide (BNP) tests. The quality of the test results was not assessed in this study.
Arm/Group | Echo, Volume Plethysmography | Brain Natriuretic Peptide (BNP)
Number analyzed (Participants) | 657 | 236
Participants | 657 | 236

2. Post Hoc Outcome: Measurement Cardiovascular Test Performance Results and Blood Flow of Left Ventricular Ejection Fraction (LVEF) and Left Ventricular Global Longitudinal Strain (GLS).
Description: An Ultrasound scan and a measurement of natriuretic peptides (BNP) in the blood were used to compute Left Ventricular Ejection Fraction (LVEF) and Left Ventricular Global Longitudinal Strain (GLS) to determine a diagnosis of Heart Failure. Theses results were compared to the results of QuantaFlo, which automatically grades the measurement results as typical for heart failure or normal. Each of the 657 participants were submitted to a brief non-invasive blood flow and cardiac performance test. A subset of 236 participants were subject to blood drawn test, Brain Natriuretic Peptide (BNP).
Time Frame: Baseline
Population: All subjects (657), adults male and female, safely had the Echo and VP tests, and after the protocol was amended, to include the Brain Natriuretic Peptide (BNP) test results of a subset of 236 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Measuring Cardiovascular Performance and Blood Flow (LVEF and GLS): Measuring cardiovascular performance and blood flow: Left Ventricular Ejection Fraction (LVEF), Ventricular Global Longitudinal Strain (GLS), was 100% safely performed for all subjects. The quality of the test results was not assessed in this study.
- Measuring Cardiovascular Performance and Blood Flow Including Brain Natriuretic Peptide (BNP).: Measure analysis when performing tests of 236 participants for Brain Natriuretic Peptide (BNP). The Protocol was amended to the data collected on 657 participants which hade Echocardiography (Echo) and Plethysmography tests.
Arm/Group | Measuring Cardiovascular Performance and Blood Flow (LVEF and GLS) | Measuring Cardiovascular Performance and Blood Flow Including Brain Natriuretic Peptide (BNP).
Number analyzed (Participants) | 657 | 236
Participants
  Male | 379 | 177
  Female | 276 | 59
  Not recorded | 2 | 0

ADVERSE EVENTS:
Time Frame: Baseline
Groups:
- Measuring Cardiovascular Performance and Blood Flow.: The feasibility of conducting all three tests on all subjects met the enrollment criteria.
Arm/Group | Measuring Cardiovascular Performance and Blood Flow.
All-Cause Mortality (participants affected / at risk) | 0/657
Serious Adverse Events (participants affected / at risk) | 0/657
Other Adverse Events (participants affected / at risk) | 0/657

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT04553484/Prot_003.pdf
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT04553484/SAP_002.pdf